CLINICAL TRIAL: NCT01446614
Title: PhaseⅠ/ⅡTrial of Autologous Bone Marrow Derived Mesenchymal Stem Cells to Patients With Parkinson's Disease.
Brief Title: Mesenchymal Stem Cells Transplantation to Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-2011-10
Record Dates: First submitted 2011-10-04; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC (Experimental): Intravenous autologous bone marrow derived mesenchymal stem cells infusion to patients with Parkinson's disease.
  Interventions: Biological: bone marrow derived mesenchymal stem cells

INTERVENTIONS:
Biological: bone marrow derived mesenchymal stem cells — Intravenous administration of up to 6x10^5 MSCs per kg,qw,for 4 weeks
  Other Names: Mesenchymal Stem Cells; Multipotent Mesenchymal Stem Cells; Multipotent Mesenchymal Stromal Cells

SUMMARY:
The study is a phase I/II trial designed to establish the safety and efficacy of intravenous administration of autologous bone marrow derived mesenchymal stem cells to patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common progressive neurodegenerative disorder caused by the loss of dopaminergic neurons in the substantia nigra. A combination of genetic and environmental factors is likely to be important in producing abnormal protein aggregation within select groups of neurones, leading to cell dysfunction and then death. A large number of agents together with surgical interventions are now available to treat early and late complications of PD, but they are suffer from two main drawbacks: side effects and loss of efficacy with disease progression.

Bone marrow (BM) derived mesenchymal stem cells (MSCs) an differentiate under certain circumstances into cells from various neuronal and glial type lineages; they also exert immunomodulatory effects. PD-derived MSCs are similar to normal MSCs in phenotype, morphology, and multidifferentiation capacity. Moreover, PD-derived MSCs are capable of differentiating into neurons in a specific medium with up to 30% having the characteristics of dopamine cells. These findings indicate that MSCs derived from PD patients' bone marrow may be a promising cell type for cellular therapy.

BM-MSCs cultured with a cocktail of growth factors (containing FGF and BDNF) differentiate into neuronal/glial lineage cells with a predominance of cells expressing astrocytes' markers. They were effective in suppression of chronic EAE in mice and induced neuroprotection, preserving most of the axons in the CNS of successfully-treated animals. Histopathological studies revealed that MSCs could efficiently migrate into the CNS inflamed tissue (both when administered intravenously and intraventricularly) and differentiated into cells expressing neural-glial lineage markers. Such an approach may provide a feasible and practical way for PD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with current diagnosis of idiopathic Parkinson's disease.
* Age 30 to 65.
* Experiencing motor complications despite optimized levodopa treatment.
* PD of Stage 2，2.5，3 or 4 of Hoehn-Yahr staging.
* Time between diagnosis and enrollment greater than 2 years.
* No significant cognitive impairment. MMSE > 24.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents within 4 weeks of study entry.
* History of allergic reactions attributed to compounds of similar biologic composition to mesenchymal stem cells.
* Primary hematologic diseases.
* Patients undergo intracranial surgeries or implantation of a device for Parkinson's disease.
* Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent and perform all study assessments.
* Atypical or secondary parkinsonism.
* Malignancy within the last 5 years.
* Any other serious medical illness that might preclude safe participation in the study.
* Pregnant or breastfeeding women.
* HIV-positive patients.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 month after transplantation

SECONDARY OUTCOMES:
Effect assessment | 1 month after transplantation
  Assessed by Unified Parkinson's Disease Rating Scale (UPDRS).
Effect assessment | 3 months after transplantation
  Assessed by UPDRS
Effect assessment | 6 months after transplantation
  Assessed by UPDRS
Effect assessment | 12 months after transplantation
  Assessed by UPDRS

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD, Study Director — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wang Y, Chen S, Yang D, Le WD. Stem cell transplantation: a promising therapy for Parkinson's disease. J Neuroimmune Pharmacol. 2007 Sep;2(3):243-50. doi: 10.1007/s11481-007-9074-2. Epub 2007 May 9. PMID 18040857
- [Background] Karussis D, Kassis I, Kurkalli BG, Slavin S. Immunomodulation and neuroprotection with mesenchymal bone marrow stem cells (MSCs): a proposed treatment for multiple sclerosis and other neuroimmunological/neurodegenerative diseases. J Neurol Sci. 2008 Feb 15;265(1-2):131-5. doi: 10.1016/j.jns.2007.05.005. Epub 2007 Jul 3. PMID 17610906
- [Background] Schwarz J, Storch A. Transplantation in Parkinson's disease: will mesenchymal stem cells help to reenter the clinical arena? Transl Res. 2010 Feb;155(2):55-6. doi: 10.1016/j.trsl.2009.08.008. Epub 2009 Sep 19. No abstract available. PMID 20129484
- [Background] Glavaski-Joksimovic A, Virag T, Mangatu TA, McGrogan M, Wang XS, Bohn MC. Glial cell line-derived neurotrophic factor-secreting genetically modified human bone marrow-derived mesenchymal stem cells promote recovery in a rat model of Parkinson's disease. J Neurosci Res. 2010 Sep;88(12):2669-81. doi: 10.1002/jnr.22435. PMID 20544825
- [Background] Somoza R, Juri C, Baes M, Wyneken U, Rubio FJ. Intranigral transplantation of epigenetically induced BDNF-secreting human mesenchymal stem cells: implications for cell-based therapies in Parkinson's disease. Biol Blood Marrow Transplant. 2010 Nov;16(11):1530-40. doi: 10.1016/j.bbmt.2010.06.006. Epub 2010 Jun 10. PMID 20542127
- [Background] Shetty P, Ravindran G, Sarang S, Thakur AM, Rao HS, Viswanathan C. Clinical grade mesenchymal stem cells transdifferentiated under xenofree conditions alleviates motor deficiencies in a rat model of Parkinson's disease. Cell Biol Int. 2009 Aug;33(8):830-8. doi: 10.1016/j.cellbi.2009.05.002. Epub 2009 May 22. PMID 19465139
- [Background] Zhang Z, Wang X, Wang S. Isolation and characterization of mesenchymal stem cells derived from bone marrow of patients with Parkinson's disease. In Vitro Cell Dev Biol Anim. 2008 May-Jun;44(5-6):169-77. doi: 10.1007/s11626-008-9093-1. Epub 2008 Apr 10. PMID 18401666
- [Background] Park HJ, Lee PH, Bang OY, Lee G, Ahn YH. Mesenchymal stem cells therapy exerts neuroprotection in a progressive animal model of Parkinson's disease. J Neurochem. 2008 Oct;107(1):141-51. doi: 10.1111/j.1471-4159.2008.05589.x. Epub 2008 Jul 28. PMID 18665911